CLINICAL TRIAL: NCT00004740
Title: Randomized Study of Interventions to Enhance Adherence to Isoniazid Prevention Therapy for Tuberculosis in Injection Drug Users
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Collaborators: Johns Hopkins University (Other)
Organization: Office of Rare Diseases (ORD) (NIH)
Allocation: Randomized | Masking: None | Purpose: Prevention
Other Study IDs: 199/11642; JHUSM-93090801
Record Dates: First submitted 2000-02-24; First posted 2000-02-25 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1998-01

CONDITIONS: Tuberculosis
Keywords: cardiovascular and respiratory diseases; rare disease; tuberculosis
MeSH Terms: conditions — Tuberculosis; Respiratory Tract Diseases; Rare Diseases | interventions — Isoniazid

INTERVENTIONS:
Drug: isoniazid

SUMMARY:
OBJECTIVES: I. Recruit 300 injection drug users with positive tuberculin skin tests who are candidates for isoniazid chemoprophylaxis into a trial of several interventions to enhance adherence to preventive therapy.

II. Compare the effectiveness of self-administered isoniazid chemoprophylaxis supplemented with peer education and support groups versus directly observed preventive therapy delivered by a licensed nurse versus self-administered therapy with standard clinic follow-up and education. Outcome measures are adherence to prescribed doses of medication and the proportion of patients who complete therapy.

III. Compare the impact of monetary incentives on therapy adherence by random assignment to immediate vs. deferred financial incentive.

IV. Assess attitudes, knowledge, and beliefs about tuberculosis and preventive therapy in these patients and determine the association of these factors with demographic, social, and clinical characteristics.

V. Assess attitudes and beliefs about tuberculosis susceptibility, seriousness, benefits of preventive therapy, barriers to therapy, and self-efficacy as predictors of health-related behaviors as measured by adherence with therapy, and determine the impact of the assigned interventions on these attitudes and beliefs.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: This is a randomized study. Patients in the first group self-administer oral isoniazid following the standard clinic protocol for 6 months. They receive individual counseling and education by a peer educator at entry and at week 2, participate in a monthly support group cofacilitated by a peer counselor and health educator, and make a monthly clinic visit.

Patients in the second group receive oral isoniazid twice a week. Therapy is administered by the nurse, who observes ingestion and swallowing. Nursing education and support per standard clinic procedures is provided at each monthly clinic visit.

Patients in the third group self-administer oral isoniazid, without enhanced education and peer support, following the standard clinic protocol for 6 months. Nursing education and support per standard clinic procedures is provided at each monthly clinic visit.

Within each group, patients are randomly assigned to an immediate or deferred financial compensation schedule. Immediate compensation for compliance with medication and clinical visit is given during the monthly clinic visit, while deferred compensation is given at study completion.

It is recommended that HIV-seropositive patients receive 6 additional months of standard isoniazid therapy.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

Population Characteristics

* Positive purified protein derivative (PPD) tuberculin skin test, with induration as follows: 10 mm or greater if HIV seronegative 5 mm or greater if HIV seropositive or status unknown
* No active tuberculosis (TB) on chest x-ray
* Candidate for isoniazid prophylaxis through Baltimore City Health Department
* Active or treated injection drug user, i.e.: Injected illicit drugs within the last 3 months OR Previously injected drugs and is in drug treatment
* Injection use documented by: Subject self report Medical and referral records from drug treatment programs Physical exam for stigmata of injection drug use

Prior/Concurrent Therapy

* No more than 6 months of prior TB preventive therapy for HIV

Subject Characteristics

* Hepatic: ALT no greater than 3 x ULN
* Renal: Not specified
* Other: No prior serious adverse reaction to isoniazid No requirement for HIV therapy other than Pneumocystis prophylaxis or antiretrovirals

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300
Dates: Start 1995-02

CONTACTS AND LOCATIONS:
Overall Officials: Richard E. Chaisson, Study Chair — Johns Hopkins University